CLINICAL TRIAL: NCT07093658
Title: Epidemiology and Outcome of High Versus Low Fall Injury in Asia Countries: A 7-year Multicenter Cohort Study
Brief Title: High vs Low Fall Injuries in Asia: 7-Year Multicenter Study
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tse-Hao Chen, Physician, Mackay Memorial Hospital
Other Study IDs: 24MMHIS447e
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Fall Injury; Trauma
Keywords: Trauma; Fall injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low fall injury group
  Interventions: Other: High fall injury group

INTERVENTIONS:
Other: High fall injury group — High fall injury group

SUMMARY:
This multicenter study revealed a declining overall incidence of fall-related injuries, accompanied by a rising proportion of high falls, predominantly among non-elderly males. Mortality risk increased significantly at fall heights of 3 and 6 meters, supporting current field triage thresholds. Across both high and low falls, lower SpO₂ and GCS were key predictors of 30-day mortality, with head injury being an additional risk factor in low fall cases

ELIGIBILITY:
Inclusion Criteria:

* This study included adult patients (aged ≥18 years) who were transported by emergency medical services (EMS) between January 2016 and December 2022.
* Fall injury patients

Exclusion Criteria:

* missing data on age, sex, injury mechanism, systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), oxygen saturation (SpO₂), Glasgow Coma Scale (GCS), Abbreviated Injury Scale (AIS) for each body region, Injury Severity Score (ISS), Revised Trauma Score (RTS), or fall height
* missing records of 30-day mortality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included adult patients (aged ≥18 years) who were transported by emergency medical services (EMS) between January 2016 and December 2022. Patients were excluded if they had missing data on age, sex, injury mechanism, systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), oxygen saturation (SpO₂), Glasgow Coma Scale (GCS), Abbreviated Injury Scale (AIS) for each body region, Injury Severity Score (ISS), Revised Trauma Score (RTS), or fall height. In addition, patients with missing records of 30-day mortality were excluded from the mortality cohort analysis.
Sampling Method: Non-Probability Sample
Enrollment: 59099 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30-day
  30-day mortality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim J, Shin SD, Im TH, Kug Jong Lee, Ko SB, Park JO, Ahn KO, Song KJ. Development and validation of the Excess Mortality Ratio-adjusted Injury Severity Score Using the International Classification of Diseases 10th Edition. Acad Emerg Med. 2009 May;16(5):454-464. doi: 10.1111/j.1553-2712.2009.00412.x. PMID 19388920
- [Background] Kong SY, Shin SD, Tanaka H, Kimura A, Song KJ, Shaun GE, Chiang WC, Kajino K, Jamaluddin SF, Wi DH, Park JO, Moon SW, Ro YS, Cone DC, Holmes JF Jr. Pan-Asian Trauma Outcomes Study (PATOS): Rationale and Methodology of an International and Multicenter Trauma Registry. Prehosp Emerg Care. 2018 Jan-Feb;22(1):58-83. doi: 10.1080/10903127.2017.1347224. Epub 2017 Aug 9. PMID 28792281